CLINICAL TRIAL: NCT05717868
Title: Effectiveness of Self-Mobilization Versus Kinesio-Taping on the Cervical Region in Electronic Device Users
Brief Title: Self-Mobilization Versus Kinesio-Taping on the Cervical Region in Electronic Device Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seth Kwame Agyenkwa, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-74555795-050.01.04-533346
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
Keywords: kinesio-taping; self-mobilization; neck disability; neck pain; electronic device users
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio-taping group (Experimental): Kinesio-tape will be applied from the dorsal region (T1-T2) to the upper cervical region (C1-C2), two times weekly in a period of four weeks.
  Interventions: Other: Kinesiology taping
- Self-mobilization group (Experimental): Self-SNAG technique will be applied by the participants with the help of a towel, and performed for a four week period.
  Interventions: Other: Self-mobilization

INTERVENTIONS:
Other: Kinesiology taping — 5 cm wide and 0.5 mm thick waterproof, porous and adhesive tape will be applied to the posterior neck of the participants while sitting comfortably in a neutral position. The first tape (Y-strip) is placed over the posterior cervical extensor muscles with approximately 25% tension. The top strip will be placed perpendicular to the Y strip on the mid-cervical region. The participant's cervical spine is flexed to obtain tension in the posterior structures.
  Arms: Kinesio-taping group
Other: Self-mobilization — The towel will be placed on the posterior arch of the fifth cervical vertebra and pulled horizontally across the face. The participant will be instructed to apply pressure to the towel and turn their head to the restricted side, then maintain the finishing interval for three seconds. The participant will be asked to apply extreme pressure in the bending position with towel support. The procedure should be painless and repeated 10 times.
  Arms: Self-mobilization group

SUMMARY:
The purpose of this clinical trial is to compare the effectiveness of kinesio-taping versus self-mobilization applied to the cervical region of long-duration electronic device users.

DETAILED DESCRIPTION:
There is increasing use of electronic devices among individuals due to technological advancement and increasing work demands. The prolong use of these devices may result to discomfort in the neck and impairments in cervical range of motion, proprioceptive sense, muscle activities, and disability among users of electronic devices. Kinesio-taping and self-mobilization in the cervical region may improve function, and reduce disability. Therefore the aim of this study is to compare the effectiveness of kinesio-taping against self-mobilization among long-duration electronic device users.

Participants will be randomized into either a kinesio-taping or self-mobilization group. Treatment will be administered within a four-week period. Participants will be evaluated at baseline, post-intervention and at one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Complain of pain in the neck
* Using electronic devices (including smart phones, desktop computers, laptops, tablets) for at least 4 hours a day,
* Using electronic devices for at least 6 months,
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of allergic reaction,
* Having previous cervical pathologies such as cervical spondylolisthesis, disc herniation, rheumatoid arthritis, muscle or ligament injury or strain,
* Having had neck or shoulder surgery,
* Having a neurological deficit (eg numbness, muscle weakness and loss of sensation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Upper trapezius electrical muscle activity | Baseline, before treatment
  The Trigno Avanti SEMG system (Delsys inc., Boston) will be used to measure the surface electromyographic activities of the upper trapezius muscle.The electrodes will be placed over the right and left trapezius muscle along the lines connecting the spinous process of the seventh cervical vertebra (C7) to the right and left acromion.
Upper trapezius electrical muscle activity | One week post-treatment (week 5)
  The Trigno Avanti SEMG system (Delsys inc., Boston) will be used to measure the surface electromyographic activities of the upper trapezius muscle.The electrodes will be placed over the right and left trapezius muscle along the lines connecting the spinous process of the seventh cervical vertebra (C7) to the right and left acromion.
Upper trapezius electrical muscle activity | One-month follow up (week 9)
  The Trigno Avanti SEMG system (Delsys inc., Boston) will be used to measure the surface electromyographic activities of the upper trapezius muscle.The electrodes will be placed over the right and left trapezius muscle along the lines connecting the spinous process of the seventh cervical vertebra (C7) to the right and left acromion.
Visaul Analogue Scale (VAS) | Baseline, before treatment
  Participants will indicate their pain level on a 10 cm horizontal line; where 0 indicates no pain and 1- the worst possible pain the subject could experience.
Visaul Analogue Scale (VAS) | One week post-treatment (week 5)
  Participants will indicate their pain level on a 10 cm horizontal line; where 0 indicates no pain and 1- the worst possible pain the subject could experience.
Visaul Analogue Scale (VAS) | One-month follow up (week 9)
  Participants will indicate their pain level on a 10 cm horizontal line; where 0 indicates no pain and 1- the worst possible pain the subject could experience.

SECONDARY OUTCOMES:
Joint Position Sense Error | Baseline, before treatment
  Joint position sense error of the cervical joint will be tested in flexion, extension, left and right rotation using a laser pointer.
Joint Position Sense Error | One week post-treatment (week 5)
  Joint position sense error of the cervical joint will be tested in flexion, extension, left and right rotation using a laser pointer.
Joint Position Sense Error | One-month follow up (week 9)
  Joint position sense error of the cervical joint will be tested in flexion, extension, left and right rotation using a laser pointer.

CONTACTS AND LOCATIONS:
Overall Officials: Rustem Mustafaoglu, Principal Investigator — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Cerrahpasa, Istanbul
  - Istanbul University-Cerrahpasa, Istanbul